CLINICAL TRIAL: NCT05133206
Title: Fasting or Non-fasting Before Cardiac Catheterization
Acronym: FORCE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Blackpool Victoria Hospital (Other)
Responsible Party: Principal Investigator, Hesham Abdelaziz, Principal Investigator, Blackpool Victoria Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 303042
Record Dates: First submitted 2021-09-09; First posted 2021-11-24 (Actual); Last update posted 2021-12-14 (Actual); Status verified 2021-12

CONDITIONS: Fasting; Coronary Artery Disease; Procedural Complication; Coronary Angiography
Keywords: Fasting; Non-fasting; Cardiac catheterization
MeSH Terms: conditions — Fasting; Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: Randomisation will take place through a sealed envelope method controlled by the cardiac research team; patients will be allocated 1:1 to either fasting or non-fasting groups using random blocks of sizes 4, 6, and 8 to minimise imbalance in treatment groups and preserve blinding up until the point of randomisation. This information (whether fasting or not) will be relayed to the patient at the time of pre-procedure assessment. The people who collate the data (the cath lab team or research nurses) and the operator performing the procedure will be blinded to the patient allocation group and will not be involved in conducting the analysis. The treatment group will be relabelled before analysis (i.e. group A and group B for not-fasting and fasting, respectively).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-Fasting (Experimental): Oral fluids and food up to the time of the procedure.
  Interventions: Other: Advice on fasting before the procedure
- Fasting (No Intervention): Clear fluids up to the time of the procedure and no food for at least 2 hours before the procedure - current practice.

INTERVENTIONS:
Other: Advice on fasting before the procedure — Patients are allowed to eat and drink freely up to the point of transfer to the Catheter Laboratory.
  Arms: Non-Fasting

SUMMARY:
The investigators hypothesise that there is no increased risk of peri-procedural complications, accompanied by improved patient satisfaction among patients allowed to eat up to the point of coronary angiography/angioplasty compared to patients, kept nil by mouth. Therefore, the investigators aim to change the practice of fasting for all patients before elective catheterization procedures.

Consented patients will be randomised in a 1:1 ratio to either fasting (standard hospital fasting policy) or non-fasting (allowed to eat and drink freely up to the point of transfer to the Catheter Laboratory).

Primary End Point will composite peri-procedural nausea, vomiting, pre-procedural hypotension, pre-procedural hypoglycemia, intra-procedural emergency endotracheal intubation and aspiration pneumonia. This will be calculated as the number of patients experiencing at least one event. Secondary end-points will include patient satisfaction questionnaire and the individual outcomes assessed in the primary end point.

DETAILED DESCRIPTION:
Nil by mouth (NBM) has been the standard of care for cardiac catheterization since its inception. The associated vomiting was common with the first generation of radiocontrast materials that were almost toxic, and with the use of general anaesthesia. Induction of anaesthesia depresses the cough and swallow reflex, thus increasing the risk of aspiration. This is also true for deep sedation. However, the practice has largely changed nowadays, with cardiac catheterization procedures being done under local anaesthesia with anxiolytic sedatives often used peri-procedurally to achieve minimal sedation whereby verbal contact is maintained. Both the Royal College of Anaesthetists and the Royal College of Emergency Medicine state that fasting is not required for minimal or conscious sedation but does recommend fasting for general anaesthesia. There is only less than a 1% risk of needing emergency surgery for percutaneous coronary interventions (PCIs). The risk of developing pulmonary aspiration following emergency coronary artery bypass grafting (CABG) surgery or emergency direct current conversion (DC) in patients without pre-procedural fasting is in the order of 0.001%.

There was no evidence that the volume or pH of participants' gastric contents differ significantly between fasting and non-fasting populations, as shown by Brady et al. In addition, the overall incidence of nausea and vomiting was reported to be 1% before elective cerebral angiography in a study carried out by Kwon et al. with no significant difference between fasting and non-fasting groups.

A recently conducted a retrospective analysis of registry data for 1916 percutaneous coronary intervention (PCI) patients over a 3-year period. None of the patients was kept nil by mouth (NBM) pre-procedure, and no patients required immediate endotracheal intubation, nor did any develop aspiration pneumonia intra or post procedurally. Thus, they concluded in their observational study that patients undergoing PCI do not need to have fasted before their procedures.

The American Society of Anaesthesia guidelines discuss this extensively and have concluded that there is no strong relation between fasting, gastric volume, or risk of aspiration. In any case, the patients at highest risk for nausea and vomiting are those who present with ST-elevation myocardial infarction (STEMI), who are not fasting anyway, and the need for emergency intubation/CABG remains rare in these patients.

Prolonged unnecessary fasting can often leave patients dissatisfied and add to the discomfort and anxiety of waiting for a procedure. Patients may also choose to miss their usual medications on the morning of the procedure due to restrictions advised with oral intake, increasing the risk of complications such as poorly controlled hypertension and the associated peri-procedural complications.

There is also evidence that patients often choose to fast longer than advised by healthcare professionals. The reasons for this include: misunderstanding by the patient that a longer period of fasting may be more protective, apprehension and loss of appetite before an invasive procedure or practical problems with timing of the procedure. Many patients undergo prolonged periods of fasting before a procedure. While this is not usually a problem for young fit patients, many of the patients do not fall into this category. Many are elderly with multiple co-morbidities and thus run the risk of hypoglycaemia and lethargy.

Further consideration has to be that of patient flow through the cardiac unit. If patients have to be NBM for a certain period before cardiac catheterization, then it reduces the ability to fill lists at short notice if patients need to be cancelled. On the other hand, if the investigators can demonstrate that this period of NBM is unnecessary, the investigators could maximize the catheter lab work as a resource.

Finally, and probably most importantly, the investigators feel that the overall patient experience will be improved if patients are allowed to eat up to the point of procedure, decreasing the number of hungry, disgruntled patients who complain to nurses.

Our pilot study of 50 patients (25 patients in each group) showed that non-fasting before cardiac catheterization is a safe and feasible approach that carries no additional risk compared to the standard practice of fasting. There was no difference in the primary composite endpoint for safety between the fasting and non-fasting group (one patient in the fasting group developed nausea/vomiting during the procedure and none in the non-fasting group; 4% vs 0, p=0.31). Compared to the fasting group, the non-fasting group had more diabetic patients (4% vs 24%, p=0.009), higher admission blood sugar (7±3 mmol/L vs 5±1 mmol/L, p=0.01), and shorter duration between the last meal and the procedure (110±85 min vs 433±158, p=009). There was no statistically significant difference between the two groups regarding the patient questionnaire results, patient satisfaction score, incidence of hypotension or chest infection within 30 days.

In summary, though growing observational evidence suggests no benefit to fasting, there is no conclusive evidence derived from a robustly randomised controlled trial to support or oppose the continued use of pre-procedural fasting before cardiac catheterisation. This proposed trial aims to add to this body of evidence and clarify guidelines and recommendations pertaining to fasting.

ELIGIBILITY:
Inclusion Criteria:

* All patients >18 years undergoing elective coronary angiography or angioplasty procedures in the 2 months window from consent.

Exclusion Criteria:

* Patients undergoing other cardiac procedures simultaneously such as EP studies, pacing and structural heart disease intervention.
* Emergency primary percutaneous coronary intervention.
* Vulnerable groups (children under 18 years old, pregnancy, mental health problems that render them unable to give informed consent).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Estimated)
Dates: Start 2022-03 (Estimated); Primary Completion 2023-08 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events as assessed by occurrence of nausea. | Within 4 hours after the procedure.
  incidence of self-reported nausea measured on a binary scale (yes or no)
Incidence of Treatment-Emergent Adverse Events as assessed by occurrence of vomiting. | Within 4 hours after the procedure.
  Incidence of vomiting assessed on binary scale (yes or no).
Incidence of Treatment-Emergent Adverse Events as assessed by occurrence of pre-procedural hypotension. | Within 2 hours before the procedure.
  Pre-procedural hypotension (systolic blood pressure <90 mmHg and /or diastolic blood pressure < 60 mmHg as measured non-invasively by sphygmomanometer)
Incidence of Treatment-Emergent Adverse Events as assessed by occurrence pre-procedural hypoglycemia. | Within 2 hours before the procedure.
  Incidence of hypoglycemia peri-procedure (blood sugar < 3.6 mmol/l) as assessed by finger prick test.
Incidence of Treatment-Emergent Adverse Events as assessed by occurrence of emergency endotracheal intubation. | During the procedure
  Incidence of emergency tracheal intubation for respiratory failure
Incidence of Treatment-Emergent Adverse Events as assessed by occurrence of aspiration pneumonia. | During the procedure
  Clinically and radiologically(X-ray and /or CT-scan) confirmed aspiration pneumonia.

SECONDARY OUTCOMES:
Patient satisfaction assessed by questionnaire using a binary score (YES or NO), qualitative assessment of free text comments and presence of other symptoms as listed in the Description | Within 4 hours after the procedure
  Questionnaire assessing the self-reported pre-procedural hunger, thirst/dry mouth, headache, weakness/lethargy, heartburn, dizziness, low mood/anxiety, ability to focus/stay mentally sharp and preferences regarding fasting on a binary scale (yes or no).

CONTACTS AND LOCATIONS:
Overall Officials: Hesham K Abdelaziz, MSc, PhD, Principal Investigator — Lancashire Cardiac Centre, Blackpool Victoria Hospital, Blackpool, United Kingdom
Locations (1):
- Blackpool Victoria Hospital, Blackpool, Lancashire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Godwin SA, Burton JH, Gerardo CJ, Hatten BW, Mace SE, Silvers SM, Fesmire FM; American College of Emergency Physicians. Clinical policy: procedural sedation and analgesia in the emergency department. Ann Emerg Med. 2014 Feb;63(2):247-58.e18. doi: 10.1016/j.annemergmed.2013.10.015. PMID 24438649
- [Background] Brady M, Kinn S, Stuart P. Preoperative fasting for adults to prevent perioperative complications. Cochrane Database Syst Rev. 2003;(4):CD004423. doi: 10.1002/14651858.CD004423. PMID 14584013
- [Background] Kwon OK, Oh CW, Park H, Bang JS, Bae HJ, Han MK, Park SH, Han MH, Kang HS, Park SK, Whang G, Kim BC, Jin SC. Is fasting necessary for elective cerebral angiography? AJNR Am J Neuroradiol. 2011 May;32(5):908-10. doi: 10.3174/ajnr.A2408. Epub 2011 Mar 17. PMID 21415144
- [Background] Hamid T, Aleem Q, Lau Y, Singh R, McDonald J, Macdonald JE, Sastry S, Arya S, Bainbridge A, Mudawi T, Balachandran K. Pre-procedural fasting for coronary interventions: is it time to change practice? Heart. 2014 Apr;100(8):658-61. doi: 10.1136/heartjnl-2013-305289. Epub 2014 Feb 12. PMID 24522621
- [Background] Practice Guidelines for Preoperative Fasting and the Use of Pharmacologic Agents to Reduce the Risk of Pulmonary Aspiration: Application to Healthy Patients Undergoing Elective Procedures: An Updated Report by the American Society of Anesthesiologists Task Force on Preoperative Fasting and the Use of Pharmacologic Agents to Reduce the Risk of Pulmonary Aspiration. Anesthesiology. 2017 Mar;126(3):376-393. doi: 10.1097/ALN.0000000000001452. No abstract available. PMID 28045707
- [Background] Naidu SS, Abbott JD, Bagai J, Blankenship J, Garcia S, Iqbal SN, Kaul P, Khuddus MA, Kirkwood L, Manoukian SV, Patel MR, Skelding K, Slotwiner D, Swaminathan RV, Welt FG, Kolansky DM. SCAI expert consensus update on best practices in the cardiac catheterization laboratory: This statement was endorsed by the American College of Cardiology (ACC), the American Heart Association (AHA), and the Heart Rhythm Society (HRS) in April 2021. Catheter Cardiovasc Interv. 2021 Aug 1;98(2):255-276. doi: 10.1002/ccd.29744. Epub 2021 May 19. PMID 33909349
- See also: Association of Anaesthetists of Great Britain and Ireland. AAGBI Safety Guideline 2010. — https://anaesthetists.org/Portals/0/PDFs/Guidelines%20PDFs/Guideline_preoperative_assessment_patient_preparation_anaesthetist_2010_final.pdf?ver=2018-07-11-163756-537&ver=2018-07-11-163756-537